CLINICAL TRIAL: NCT05318196
Title: Molecular Prediction of Development, Progression or Complications of Kidney, Immune or Transplantation-related Diseases
Acronym: NEPHROGENE2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0154
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury; Chronic Kidney Diseases; Solid-organ Transplantation; Cancer; Metabolic Disease; Immune Diseases
Keywords: risk stratification; solid-organ transplantation; cancer; Chronic kidney disease; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Neoplasms; Metabolic Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Biological samples collection — SOT patients: samples will be collected at the time of the protocol follow-up visit (registration on the transplant list, on the day of the transplantation, and then at day 15, month 1-3-6-9-12 and then annually, as well as if complications or therapeutic modifications).
  Dialysis patients: at the start of the dialysis and then at M3, M12, and if complications or modification of the dialysis protocol.
  Non-dialysis or cancer patients: the sampling frequency will be individualized according to the pathology studied (acute or chronic) and the purpose of the sampling (diagnostic, mechanistic, prediction, evaluation of the therapeutic response). Samples for diagnostic and mechanistic purposes will be taken only once. Samples for prognostic purposes will be taken at regular intervals, adapted to the natural history of the disease while respecting the maximum volume of blood samples defined by the French law. Samples will be collected during a sampling performed as part of routine care.

SUMMARY:
Managing patients with renal failure requires an understanding of the molecular mechanisms that lead to its occurrence (i.e. upstream of the disease), its worsening and its persistence (i.e. downstream), while also specifying the risk of worsening renal failure (risk stratification, intolerance to the treatment or complications (infectious, metabolic, cardiovascular, cancer…). Nephrogene 2.0 aims to study these different components of kidney, immune and solid organ transplantation (SOT)-related diseases.

DETAILED DESCRIPTION:
Acute renal failure (ARF) and chronic kidney disease (CKD) are frequent pathologies (850 million people are affected worldwide). Renal failure is associated with an increased morbidity and mortality, including an increased risk of infections, drug toxicity and cardiovascular death. The causes of renal failure are numerous: metabolic (diabetes, hypertension), immunological (autoimmune diseases, monoclonal gammopathies), toxic (environment, drugs), genetic, infectious, ischemic, paraneoplastic... Any episode of ARF is also accompanied by a risk of secondary CKD (relative risk multiplied by 9).

The mechanisms leading to renal failure are multiple and combine predisposing genetic factors, inadequate intra-renal or systemic immune response, endothelial and epithelial dysfunctions, and potentially inappropriate regenerative capacity. In addition, renal failure or its treatment itself may be accompanied by additional renal lesions (e.g. nephrotoxicity of calcineurin inhibitors used as anti-rejection treatment in transplantation, hemodynamic intolerance with secondary ARF during hemodialysis sessions, iatrogenic ARF when using diuretics or inhibitors of the renin angiotensin system) or extra-renal complications (e.g. immunosuppression and infections induced by immunomodulatory therapies during autoimmune diseases or for prevention of transplant rejection; vascular diseases secondary to phosphocalcic disorders).

Patients included in the NEPHROGENE 2.0 cohort will be followed during 10 years and clinical data and biological samples will be collected at the inclusion in the cohort, at each monitoring programmed in their usual care and and at each event (infection, acute kidney injury, cancer…). Samples will be collected according to the symptoms of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (> 18 year of age) with kidney disease or at risk to develop a kidney disease,
* Patients followed by a practitioner of the Department of Nephrology and Organ Transplantations of the University Hospital of Toulouse (France)

Exclusion Criteria:

* consent deny
* inability of the patient or its family to give consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who develop or have progression of kidney, immune or transplantation-related diseases, as well as specific complications of these conditions
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Identification of the molecular mechanisms underlying kidney, immune and solid organ transplantation-related diseases. | yearly and up to 10 years after inclusion in the study
  To identify the molecular mechanisms underlying kidney, immune and solid organ transplantation-related diseases. An unbiased multi-omic approach (including peptidomics, metabolomics, genome sequencing, and flow cytometry and transcriptomic of circulating immune cells) will be performed at the inclusion in the study and correlated to specific end-points (acute kidney injury, kidney failure progression, end-stage kidney disease, infection, cancer according to the underlying condition). Multiple measurements will be studied individually to identify genes variations, gene expression changes, urinary or plasma peptides abundance, immune cells relative abundance in the blood that correlate with the end-point. In a second step, an attempt to combine them in a single predictive signature using artificial intelligence approach.

SECONDARY OUTCOMES:
Identification of the predictive factors (immunological, metabolic, genetic…) for the development or progression of renal diseases | up to 10 years after inclusion in the study
  To identify the predictive factors (immunological, metabolic, genetic…) for the development or progression of renal diseases: end-points will be end-stage kidney disease, or a decrease of the estimated glomerular filtration rate (eGFR) > 50%
Identification of the molecular mechanisms (immunological, genetic…) driving complications of kidney, immune and SOT-related diseases | up to 10 years after inclusion in the study
  To identify the molecular mechanisms (immunological, genetic…) driving complications of kidney, immune and SOT-related diseases: end-points will the development of bacterial, viral (CytoMégaloVirus, Herpes simplex virus, varicella-zoster virus, BK virus…) or fungal (candidiasis, aspergillosis…) infections, as well as cardiovascular events or other complications
To specify the individual risk of complications secondary to SOT or its treatment | up to 10 years after inclusion in the study
  To specify the individual risk of renal and immunological complications secondary to cancer or hematological malignancies, or their treatments: end points will be the development of acute kidney injury, end-stage kidney disease or >50% reduction of the eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Faguer, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Rangueil University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No